CLINICAL TRIAL: NCT01577849
Title: Randomized, Open-label Crossover Study to Evaluate Comparative Pharmacokinetics of Vitamin D3 Between DP-R206(150mg Ibandronate / 24,000 IU Vitamin D3 Tablet) and a 24,000 IU Vitamin D3 in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetic Characteristics of DP-R206(Vitamin D3) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DP-CTR206-02
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
MeSH Terms: interventions — Cholecalciferol; DP-R206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Active Comparator)
  Interventions: Drug: Vitamin D3
- DP-R206 (Experimental)
  Interventions: Drug: DP-R206

INTERVENTIONS:
Drug: Vitamin D3 — administration of Vitamin D3 24,000 IU
  Arms: Vitamin D3
Drug: DP-R206 — administration of DP-R206 (150mg ibandronate / 24,000IU Vitamin D3)
  Arms: DP-R206

SUMMARY:
The purpose of this study is to compare the pharmacokinetic characteristics of DP-R206 (150mg Ibandronate / 24,000 IU Vitamin D3 complex tablet, qd) and Vitamin D3 (24,000 IU Vitamin D3 , qd) after oral administration in healthy adult volunteers.

DETAILED DESCRIPTION:
The number of patient is thirty-six. Patients were randomly assigned either a Vitamin D3 tablet(24,000 IU Vitamin D3, qd) first, DP-R206(150mg Ibandronate / 24,000 IU Vitamin D3 complex tablet, qd) Second or DP-R206(150mg Ibandronate / 24,000 IU Vitamin D3 complex tablet, qd) first, Vitamin D3 tablet(24,000 IU Vitamin D3 , qd) second.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of healthy volunteers

Exclusion Criteria:

* Hypersensitivity Reaction about Ibandronate or other drugs(aspirin, antibiotics)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetics | 24, -18, -12, -6, 0(predose), 1, 4, 6, 8, 10, 16, 24, 36, 48, 72, 96, 120 hours post-dose
  Cmax, AUClast

SECONDARY OUTCOMES:
Composite of pharmacokinetics | 24, -18, -12, -6, 0(predose), 1, 4, 6, 8, 10, 16, 24, 36, 48, 72, 96, 120 hours post-dose
  AUCinf, tmax, t½β

CONTACTS AND LOCATIONS:
Overall Officials: Min Gul KIM, MD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk national University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Jeon JY, Lee SY, Im YJ, Kim EY, Kim Y, Park TS, Chae SW, Lee JW, Jun H, Lee TW, Kim MG. Comparison of the pharmacokinetics, safety, and tolerability of vitamin D3 in DP-R206 (150-mg ibandronate/24,000-IU vitamin D3 tablet) and as monotherapy (24,000 iu) in healthy male Korean adults. Clin Ther. 2014 Jan 1;36(1):48-57. doi: 10.1016/j.clinthera.2013.12.001. Epub 2013 Dec 28. PMID 24378207